CLINICAL TRIAL: NCT03170115
Title: Phase II Randomized Study of Induction Chemotherapy Followed by Chemoradiotherapy With or Without Aspirin in High Risk Locally Advanced Rectal Cancer
Brief Title: Induction Chemotherapy Plus Chemoradiotherapy With or Without Aspirin in High Risk Rectal Cancer
Acronym: ICAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Aspirin added to chemoradiotherapy was safe but did not improve response to total neoadjuvant treatment. The study was closed due absence of benefit.
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICAR trial
Record Dates: First submitted 2017-04-17; First posted 2017-05-30 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Rectal Cancer, Adenocarcinoma; Locally Advanced Malignant Neoplasm; Chemoradiation
Keywords: Rectal Cancer; Total neoadjuvant therapy; Induction chemotherapy; Aspirin colorectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Aspirin; N-hydroxy-4-acetylaminostilbene

STUDY DESIGN:
Intervention Model Description: preoperative induction chemotherapy followed by combined radiochemotherapy with capecitabine and aspirin
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aspirin (Experimental): Induction chemotherapy followed by chemoradiotherapy with aspirin Aspirin 100mg daily during the chemoradiotherapy
  Interventions: Drug: Aspirin
- Placebo Oral Tablet (Placebo Comparator): Induction chemotherapy followed by chemoradiotherapy without aspirin Placebo daily during the chemoradiotherapy
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Aspirin — chemoradiotherapy with capecitabine and aspirin Aspirin daily during chemoradiotherapy
  Other Names: aas
  Arms: Aspirin
Drug: Placebo Oral Tablet — chemoradiotherapy with capecitabine and placebo Placebo daily during chemoradiotherapy
  Other Names: placebo
  Arms: Placebo Oral Tablet

SUMMARY:
The benefit of aspirin in cancer of the colon and rectum is already known. Recently, it was described its potential activity during chemoradiotherapy, with higher rate of tumor downstaging. Furthermore, induction chemotherapy followed by chemoradiation represents an attractive approach, with more favorable compliance and toxicity profiles. The aim of this study was to evaluate the efficacy of total neoadjuvant treatment and assess the efficacy and feasibility of aspirin use during chemoradiotherapy for high-risk rectal cancer.

DETAILED DESCRIPTION:
Methods: This is a randomized trial to evaluate induction treatment with XELOX and Capecitabine-based chemoradiotherapy with or without aspirin in a high-risk population selected by MRI. High-risk will be defined by presence of at least one of the following criteria on high-resolution thin-slice MRI (3 mm): tumors extending to within 1 mm of, or beyond the mesorectal fascia; tumor extending 5 mm or more into perirectal fat; resectable cT4 tumors; lower third; nodal involvement; extramural vascular invasion. Random assignment of treatment will be stratified by MRI tumour regression grade. All the patients enrolled in the study will receive XELOX every 21 days for four cycles, unless unacceptable toxicity or progression is detected. After this treatment, patients will be randomized to receive Capecitabine-based chemoradiotherapy with aspirin or placebo (Capecitabine 850 mg/m² 5 days per week combined with radiotherapy with total dose of 50.4 Gy in 28 days). After 8-10 weeks, they will be evaluate by MRI. Patients with incomplete clinical response will be referred to immediate surgery and patients with complete clinical response will be managed with "watch and wait" approach. Patients with progression disease during the treatment phase will be withdrawn from the study and will receive their treatment according to the investigator's judgment.

The sample size was calculated according to Simon's optimal two-stage design. Accordingly, 11 patients must be included in each group during the first stage and 20 during the second stage. A treatment regimen will be considered effective if more than 18 patients of the total 31 show downstaging (final analysis), reaching 80% power with an alpha of 0.05 level of significance.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of mid or low rectum
2. Locally advanced rectal cancer with one of the high-risk factors confirmed by high-resolution thin-slice Magnetic resonance image (3 mm)

   * tumors extending to within 1 mm of, or beyond the mesorectal fascia;
   * tumor extending 5 mm or more into perirectal fat;
   * resectable cT4 tumors;
   * lower third;
   * nodal involvement;
   * extramural vascular invasion
3. ECOG performance status of 0-2
4. An informed consent has been signed by the patient

Exclusion Criteria:

1. Upper rectal cancer
2. Metastatic disease
3. The patient received any previous therapy for colorectal cancer or another malignancy
4. Other malignant tumours within the last 5 years except cervical carcinoma in situ and basal cell carcinoma of the skin
5. Previous thromboembolic or haemorrhagic events within 6 months prior to registration
6. Patients with malabsorption syndrome or difficulties in swallowing
7. The patient has severe underlying diseases or poor condition to receive chemotherapy or radiotherapy
8. Pregnant of breastfeeding women
9. The patient who participate in another clinical trial, or receives any drug for the trial
10. Uncontrolled peripheral neuropathy (more than grade 2)
11. Active gastrointestinal bleeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Tumor downstaging after induction chemotherapy followed by chemoradiotherapy with or without aspirin | 8-10 weeks after chemoradiotherapy
  This will be assessed by MR imaging 8-10 weeks after chemoradiotherapy and it will be considered tumor downstaging if mrTRG 1 to 3

SECONDARY OUTCOMES:
Radiological Tumor response rate after induction chemotherapy | 3-4 weeks after last induction chemotherapy
  This will be assessed by MR imaging after induction chemotherapy
Pathological Tumor response rate | 10-12 weeks after chemoradiotherapy
  Amount of tumor regression after surgery according to the guideline including Mandard
Pathologic complete response | 8-10 weeks after chemoradiotherapy
  it will be defined as the absence of residual invasive cancer on pathological evaluation of the complete resected rectal specimen
Disease-free survival | 3 years
  defined as the time from surgery to relapse or death, whichever occurred first
Overall survival | 5 years
  defined as the time from surgery to death, whichever occurred first

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Henrique Araujo, MD, PHD, Principal Investigator — National Cancer Institute, France
Locations (1):
- INCA- Instituto Nacional de Câncer, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No